CLINICAL TRIAL: NCT00373971
Title: Nutritional Care - Preventing Loss of Weight, Fat Free Mass and Activities of Daily Living Four Months After Surgery.
Brief Title: Preventing Loss of Weight, Fat Free Mass and Activities of Daily Living
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Allocation: Non-Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 1995-1-62
Record Dates: First submitted 2006-09-07; First posted 2006-09-08 (Estimated); Last update posted 2006-09-08 (Estimated); Status verified 2006-09

CONDITIONS: Hip Fracture; Arthrosis
Keywords: Activities of daily living; Elderly; Nutrition; Postoperative; Hip fractures; Hip replacement; Knee replacement
MeSH Terms: conditions — Hip Fractures; Osteoarthritis

INTERVENTIONS:
Behavioral: Involving the patients in their own nutritional care

SUMMARY:
Malnutrition of elder orthopaedic patients leads to weight loss and loss of fat free mass. Changes in the individual's nutritional status and body composition may adversely affect the patient's postoperative level of activity.

Aim. Thus, the purpose of the present study is to report changes in postoperative weight, FFM and functions vital to daily living in a group of elder orthopaedic patients that were actively involved in their nutritional care during the hospital stay.

DETAILED DESCRIPTION:
Malnutrition of elder orthopaedic patients leads to weight loss and loss of fat free mass. Changes in the individual's nutritional status and body composition may adversely affect the patient's postoperative level of activity.

Aim. Thus, the purpose of the present study is to report changes in postoperative weight, FFM and functions vital to daily living in a group of elder orthopaedic patients that were actively involved in their nutritional care during the hospital stay.

Method. The study comprises 253 patients aged 65+ and admitted either for hip- or knee replacement or with a fractured hip. Following a quasi-experimental design, 142 patients were allocated to the control group and 109 patients to the intervention group. The intervention programme focused on patients' involvement in their nutritional care. Body composition by bio impedance and functional status by a standard chart were assessed at admission and four months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 and above admitted either for elective hip- or knee replacement or acute with a fractured hip were allocated to the study. Patients included in the study were to stay in hospital for more than 7 days and agree on coming to the outpatient clinic for a follow-up four months after surgery.

Exclusion Criteria:

* Patients who refused to participate, patients were not able to understand the instructions,or received dietary treatment due to DM. Patients who suffered from cancer, gastrointestinal disorders or were undergoing steroid treatment. In addition, patients who were unable to participate due to serious heart disorders; or were transferred to intensive or cardiac units after surgery and did not return to the ward.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 252
Dates: Start 1995-11; Study Completion 1998-07

PRIMARY OUTCOMES:
Changes in weight
Changes in Fatt Free Mass
Changes in ADL-activities

SECONDARY OUTCOMES:
energy intake
Protein intake

CONTACTS AND LOCATIONS:
Overall Officials: Preben U Pedersen, phd, Principal Investigator
Locations (1):
- County hopital of Koge, Køge, Denmark